CLINICAL TRIAL: NCT05098743
Title: The Influence of a Medication Adherence Smartphone Application on Medication Adherence in Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Christa Hartch, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 211409
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Medication Adherence; Self Efficacy
Keywords: Medication Knowledge; Medication Social Support; Medication Self Efficacy; Mobile Phone Applications; Medically Underserved Populations
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants using the medication adherence mobile application. (Experimental): Participants in this arm will use the Medisafe app to receive medication reminders for thirty days.
  Interventions: Behavioral: Medisafe smartphone mobile application
- Participants using a printed copy of their medication list. (Active Comparator): Participants in this arm will use a printed out copy of their medication list for thirty days.
  Interventions: Behavioral: Printed medication list

INTERVENTIONS:
Behavioral: Medisafe smartphone mobile application — The medication adherence smartphone mobile application (app) will provide reminders to take individual patient medications and offers medication information and a social support feature.
  Arms: Participants using the medication adherence mobile application.
Behavioral: Printed medication list — Patients will receive a printed out medication list from their electronic medical record.
  Arms: Participants using a printed copy of their medication list.

SUMMARY:
Medication adherence is a critical aspect of achieving optimal health outcomes. Thirty to 50% of patients adhere to long-term medication treatment of chronic diseases. Non adherence has been shown to result in worsening disease, increased healthcare expenditures, complications and even death. Medically underserved communities have higher rates of medication nonadherence and a higher prevalence of chronic conditions and often receive care at Federally Qualified Health Centers (FQHCs) which are reporting caring for increasingly complex chronic conditions. Smartphone mobile phone ownership has increased to 76% in low income Americans, but this population has been underrepresented in mobile health intervention studies. This two-group, cluster randomized by site, randomized controlled trial will investigate the effect of a medication adherence smartphone mobile application (app) which provides reminders on patient medication adherence, on medication self-efficacy, medication knowledge and medication social support. Independently, each of these concepts have been shown to support medication adherence. However in the context of delivery by a medication adherence app in a variety of chronic illnesses in a medically underserved population, little is known. It will also explore if those who accessed educational materials within the app report greater medication knowledge than those who do not and if participants who choose to use the additional Medfriend feature report greater medication social support than those who do not. The study will also explore patients' perceptions on the usefulness and satisfaction with the app features.

DETAILED DESCRIPTION:
Medication adherence is a critical aspect of achieving optimal health outcomes. Thirty to 50% of patients adhere to long-term medication treatment of chronic diseases. Non adherence has been shown to result in worsening disease, increased healthcare expenditures, complications and even death. Medically underserved communities have higher rates of medication nonadherence and a higher prevalence of chronic conditions and often receive care at Federally Qualified Health Centers (FQHCs) which are reporting caring for increasingly complex chronic conditions. Smartphone mobile phone ownership has increased to 76% in low income Americans, but this population has been underrepresented in mobile health intervention studies. This two-group, cluster randomized by site, randomized controlled trial will investigate the effect of a medication adherence smartphone mobile application (app) which provides reminders on patient medication adherence, on medication self-efficacy, medication knowledge and medication social support. Independently, each of these concepts have been shown to support medication adherence. However in the context of delivery by a medication adherence app in a variety of chronic illnesses in a medically underserved population, little is known. It will also explore if those who accessed educational materials within the app report greater medication knowledge than those who do not and if participants who choose to use the additional Medfriend feature report greater medication social support than those who do not. The study will also explore patients' perceptions on the usefulness and satisfaction with the app features.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years and older
* speak and understand English
* personally own and use an Android or Apple smartphone and
* take at least 1 medication for a chronic illness based on their computerized medical record at the health center.

Exclusion Criteria:

* already using a medication reminder app or other electronic reminder system such as phone alarms
* own smartphones that are not capable of downloading the app
* patients with severe dementia or serious mental illness, and
* inability to use a mobile phone or the medication reminder software either physically or cognitively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deonni P Stolldorf, PhD, RN, Study Chair — Vanderbilt University
Locations (2):
- United States (2):
  - NCHC's Smilow Life Center, Norwalk, Connecticut
  - Norwalk Community Health Center, Inc. (NCHC), Norwalk, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartch C, Dietrich MS, Lancaster BJ, Mulvaney SA, Stolldorf DP. Satisfaction and Usability of a Commercially Available Medication Adherence App (Medisafe) Among Medically Underserved Patients With Chronic Illnesses: Survey Study. JMIR Hum Factors. 2025 Jan 7;12:e63653. doi: 10.2196/63653. PMID 39773694
- [Derived] Hartch CE, Dietrich MS, Lancaster BJ, Stolldorf DP, Mulvaney SA. Effects of a medication adherence app among medically underserved adults with chronic illness: a randomized controlled trial. J Behav Med. 2024 Jun;47(3):389-404. doi: 10.1007/s10865-023-00446-2. Epub 2023 Dec 21. PMID 38127174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a healthcare center, as noted in the protocol section.
Period: Overall Study
Arm/Group | Participants Using the Medication Adherence Mobile Application. | Participants Using a Printed Copy of Their Medication List.
Started | 32 | 33
Completed | 30 | 31
Not Completed | 2 | 2
Not completed — One participant had no data because they were unable to download the app despite multiple attempts | 1 | 0
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Using the Medication Adherence Mobile Application. | Participants Using a Printed Copy of Their Medication List. | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 25 | 52
  >=65 years | 3 | 6 | 9
Age, Continuous [Median (Full Range); unit: years] | 53.50 [37 to 76] | 51 [21 to 76] | 53 [21 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 13 | 19 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5 | 2 | 7
  Black or African American | 10 | 13 | 23
  Hispanic/Latino | 4 | 10 | 14
  Native American or Alaska Native | 1 | 0 | 1
  White | 6 | 3 | 9
  Other | 3 | 2 | 5
  Chose not to respond | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 31 | 61
ARMS [Median (Inter-Quartile Range); unit: units on a scale] | 18.5 [14 to 25] | 17.0 [14 to 21] | 18.0 [14.5 to 21.5]
SEAMS [Median (Inter-Quartile Range); unit: units on a scale] | 29.0 [25 to 36] | 31.0 [26 to 39] | 29.0 [26.0 to 38.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Medication Adherence as Measured by the Adherence to Refills and Medications Scale (ARMS)
Description: The ARMS is a global (continuous) 12-item scale, responses range from 1 (none) to 4 (all of the time) with a possible score of 12-48, patients with low ARMS scores indicate better adherence, it is valid and reliable in a low-literacy chronic disease population.
Time Frame: Baseline to 30 days.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Participants Using the Medication Adherence Mobile Application. | Participants Using a Printed Copy of Their Medication List.
Number analyzed (Participants) | 30 | 31
score on a scale | -4.0 [-8 to -1] | -1.0 [-3 to 0]

2. Primary Outcome: Change in Medication Self-efficacy as Measured by the Self-efficacy for Appropriate Medication Use Scale (SEAMS)
Description: The SEAMS is a global (continuous) 13-item scale, responses range from 1 (not confident) to 3 (very confident), with a possible score of 13-39. Patients with higher scores indicate higher levels of self-efficacy for medication adherence. It is valid and reliable in low-literacy chronic disease populations. Patients are asked their level of confidence about taking medications correctly.
Time Frame: Baseline to 30 days.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Participants Using the Medication Adherence Mobile Application. | Participants Using a Printed Copy of Their Medication List.
Number analyzed (Participants) | 30 | 31
score on a scale | 3.5 [0 to 8] | 0.0 [-3 to 3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through enrollment to study completion, an average of 30 days for each participant.
Description: There were no adverse events reported through study completion, an average of 30 days for each participant.
Arm/Group | Participants Using the Medication Adherence Mobile Application. | Participants Using a Printed Copy of Their Medication List.
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT05098743/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT05098743/ICF_001.pdf